CLINICAL TRIAL: NCT05148754
Title: An Open-label Clinical Study of the Pharmacokinetics and Safety of Elsulfavirine, 200 mg Tablets, With Single and Multiple Oral Administration in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COVID-VM1500-02
Record Dates: First submitted 2021-12-06; First posted 2021-12-08 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-02

CONDITIONS: Covid19; HIV-1-infection
Keywords: Elsulfavirine; HIV-1; 2019-nCoV; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — elsulfavirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Elsulfavirin 400 mg. (Experimental): Cohort I (N = 3). Single oral dose of 400 mg.
  Interventions: Drug: Elsulfavirine
- Elsulfavirin 800 mg. (Experimental): Cohort II (N = 3). Single oral dose of 800 mg.
  Interventions: Drug: Elsulfavirine
- Elsulfavirin 1 200 mg. (Experimental): Cohort III (N = 3). Single oral administration at a dose of 1200 mg.
  Interventions: Drug: Elsulfavirine
- Elsulfavirin 1 200 mg*9 (Experimental): Cohort IV (N = 6). A single 1200 mg oral dose followed by 200 mg daily for 9 days.
  Interventions: Drug: Elsulfavirine

INTERVENTIONS:
Drug: Elsulfavirine — Elsulfavirin 200 mg tablets.
  Other Names: VM-1500

SUMMARY:
An open-label clinical study of the pharmacokinetics and safety of Elsulfavirine, 200 mg tablets, with single and multiple oral administration in healthy volunteers.

DETAILED DESCRIPTION:
The present study is an open-label, single-center, clinical study of the pharmacokinetics and safety of Elsulfavirin 200 mg tablets in four dosage regimens:

* Cohort I (N = 3). Single oral dose of 400 mg.
* Cohort II (N = 3). Single oral dose of 800 mg.
* Cohort III (N = 3). Single oral administration at a dose of 1200 mg.
* Cohort IV (N = 6). A single 1200 mg oral dose followed by 200 mg daily for 9 days.

The study is descriptive and will not test any hypotheses. Based on previous studies and the intended descriptive objectives of the study, no control group is planned.

To ensure safety, the following scheme for using the investigational drug is provided:

* The inclusion in the study of volunteers included in each subsequent cohort will be carried out strictly after the completion of the study by the last study subject included in the previous cohort and obtaining a safety opinion.
* Dosing in the multiple administration cohort will be 2 + 4. Initially, 2 volunteers will be included, after completion of participation, 4 more volunteers will be dosed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female between the ages of 18 and 45 years (inclusive).
2. Body mass index in the range of 18.6-29.9 kg / m 2 inclusive;
3. Verified diagnosis medically fit according to the data from standard clinical, laboratory and instrumental examination methods;
4. Systolic blood pressure is not less than 100 mm hg and not higher than 130 mm hg ; diastolic blood pressure not less than 60 mm hg and not higher than 90 mm hg; pulse rate not less than 60 beats / min and not more than 90 beats / min, respiratory rate within 12-20 per minute; body temperature not less than 35.9 ° С and not more than 36.9 ° С.
5. The ability to understand and comprehend the explanation about the research;
6. Willingness to comply with all procedures and restrictions associated with research;
7. The written informed consent of the volunteer to participate in the study in accordance with the current legislation, obtained before the start of any research procedures;
8. For women with preserved reproductive potential - a negative pregnancy test and consent to adhere to adequate contraceptive methods from the screening visit up to 180 days after the last intake of the study drug, inclusively, or lack of reproductive potential;
9. For men - consent to adhere to adequate contraceptive methods with partners with preserved reproductive potential from the first day of screening to 180 days after the last dose of the study drug, inclusive.

Exclusion Criteria:

A volunteer will not be included in the study if at least one of the following criteria is met:

1. Drug intolerance to any drug;
2. Relevant history of allergies
3. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
4. Acute infectious diseases or allergic reactions requiring treatment (including drug allergies) less than 4 weeks before the first day of screening;
5. Surgical interventions on the gastrointestinal tract (except appendectomy);
6. Volunteers with suspected hypersensitivity to study drugs or any of their components;
7. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood or other conditions that make it impossible for a volunteer to participate in the study, according to the researcher;
8. The results of standard laboratory and instrumental examination tests obtained during the screening, which go beyond the normal values;
9. A positive result for at least one of the following tests:
10. blood test for HIV;
11. blood test for Syphilis;
12. blood test for hepatitis B;
13. blood test for hepatitis C;
14. Positive AOB results;
15. Positive results of urine test for the content of narcotic and potent substances;
16. Positive urine pregnancy test results in female volunteers;
17. Any diet, such as a vegetarian diet, within 2 weeks of the first day of screening;
18. Reception of more than 10 units. alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml of wine or 50 ml of strong alcoholic beverages) or history of alcoholism, drug addiction, drug abuse;
19. Inability to go without food for at least 12 hours and inability to take the drug on an empty stomach;
20. Donation of blood (450 ml of blood or plasma and more) less than 3 months before the first day of screening;
21. Depot injections, installation of intrauterine hormonal therapeutic systems or implants of any drugs 6 months before the first day of screening;
22. For females: use of hormonal contraceptives less than 2 months before the first day of screening;
23. Regular medicinal drug intake less than 2 weeks before the first day of screening;
24. Taking medications that have a pronounced effect on hemodynamics, the function of liver microsomal enzymes, the function of the gastrointestinal tract, etc. (barbiturates, omeprazole, cimetidine, etc.), vitamins and or dietary supplements less than 30 days before the first day of screening;
25. For females: volunteers with preserved reproductive potential who had unprotected intercourse with an unsterilized male partner within 30 days before the first day of screening;
26. For females: Breast-feeding period
27. Participation in any other clinical trial or study drug intake less than 3 months before the first day of screening;
28. Difficulty accessing a vein, making it difficult or impossible to insert a catheter and perform a frequent blood sampling;
29. Smoking.
30. Volunteers unwilling or unable to give up alcohol and excessive exercise from the first day of screening to the follow-up visit;
31. Volunteers who are unwilling or unable to avoid food and drinks containing methylxanthines and grapefruit / grapefruit juice from the first day of screening to the follow-up visit;
32. Volunteers with lifestyles (including night work and extreme physical activity such as sports or weight lifting) that can make it difficult to interpret laboratory findings from the study;
33. Volunteers who do not intend to comply with the research regime and / or are not credible to the researcher;
34. Volunteers who are clearly or likely, in the opinion of the researcher, are not able to understand and evaluate the information on this research as part of the informed consent form signing process, in particular regarding the expected risks and possible discomfort;
35. Dehydration due to diarrhea, vomiting or other reason within the last 24 hours before the first day of screening;
36. A history of seizures, epilepsy and any other neurological disorders;

Criteria of exclusion (withdrawn of a volunteer from the study at the initiative of the researcher):

1. The researcher decided that the volunteer should be excluded in the interests of the volunteer;
2. Non-compliance with the exclusion criteria identified during the study. Deviations of indicators of vital body functions, as well as standard laboratory and instrumental indicators from the established normal values, detected after the volunteer took the study drug, are considered an undesirable phenomenon;
3. The occurrence of AEs / SAEs when the continuation of the volunteer's participation in the study is undesirable or impossible (according to the sponsor / manufacturer or researcher);
4. Vomiting or diarrhea within 8 hours after taking the drug;
5. Unauthorized concomitant treatment (protocol violation);
6. Non-compliance by the volunteer with the rules of stay at the clinical base;
7. The volunteer is receiving additional treatment (or needs additional treatment, including the use of additional drugs) that may affect the pharmacokinetics of the study drugs;
8. The volunteer requires inpatient treatment during the study;
9. Volunteers arrive at the hospital later than the appointed time (more than 1 hour late), which violates the protocol requirements;
10. Positive AOB results;
11. Positive pregnancy test;
12. Positive results of urine test for the content of narcotic and potent substances;
13. In the adverse events that the resulting side effects of the drug are so serious that continuation of the study is unacceptable.

The expulsion of the volunteer at the initiative of the researcher.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of Elsulfavirine, 200 mg tablets, in healthy volunteers. The incidence of AEs and SAEs. | Cohort I-III Not more than 28 days. Cohort IV Not more than 39 days.
  To evaluate the pharmacokinetics of Elsulfavirine, 200 mg tablets, in healthy volunteers. Describe and study the pharmacokinetic parameters and relative bioavailability of the study drug for different modes of administration. Conduct an assessment and comparative analysis of the safety and tolerability of the study drug based on data on adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Rodyukova, PhD, Principal Investigator — V. P. Demikhov City Clinical Hospital of the Department of Healthcare of the City of Moscow
Locations (1):
- State Budgetary Institution Healthcare of the City of Moscow " V. P. Demikhov City Clinical Hospital of the Department of Healthcare of the City of Moscow", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No